CLINICAL TRIAL: NCT01325948
Title: Cross-sectional Observational Study to Investigate the Effects of Chronic Obstructive Pulmonary Disease on Daily Life Activities
Brief Title: Cross-sectional Study to Investigate the Effects of Chronic Obstructive Pulmonary Disease on Daily Life Activities
Acronym: COPD LIFE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Mujgan Ates / MC MD, AstraZeneca
Other Study IDs: NIS-RTR-XXX-2011/1
Record Dates: First submitted 2011-03-21; First posted 2011-03-30 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with COPD

SUMMARY:
The purpose of this study is to investigate the effects of Chronic Obstructive Pulmonary Disease (COPD) on daily life activities in patients with COPD and also to determine the socio-demographic profile, daily life style and needs of the patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Outpatient treatment for any reason
* Current or ex-smoker

Exclusion Criteria:

* An exacerbation of COPD that still lasts or that was experienced within last 3 months
* History of asthma and/or allergic rhinitis
* The presence of another important respiratory disease

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from health institutions where the patients with COPD are treated
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Effect of COPD on daily activities | 1 year
  The distribution of the patients according to their answers, as Yes / No / Unknown, given to the questions of patient questionnaire about the effect of COPD on daily life and which daily activities are limited will be calculated as percentage.

SECONDARY OUTCOMES:
Patients' socio-demographic profiles, daily life conditions and needs and expectations from therapy | Baseline
  The answers the patients give to the questions about socio-demographic profiles, daily life conditions and needs and their expectations from the therapy will be summarized as percentages: Age and gender, educational background, place of residence, marital status and life conditions, concomitant diseases, smoking status, the diagnosis of COPD and its clinical characteristics basic knowledge of the patient about COPD daily life of the patient, expectations from the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Goztas, Study Director — AstraZeneca Turkey; Mehmet Polatli, Principal Investigator — Adnan Menderes University Faculty of Medicine
Locations (20):
- Turkey (Türkiye) (20):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Aydin
  - Research Site, Bartın
  - Research Site, Bolu
  - Research Site, Burdur
  - Research Site, Bursa
  - Research Site, Gaziantep
  - Research Site, Gebze
  - Research Site, Giresun
  - Research Site, Isparta
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Karabük
  - Research Site, Kayseri
  - Research Site, Konya
  - Research Site, Manisa
  - Research Site, Mersin
  - Research Site, Yozgat